CLINICAL TRIAL: NCT07384780
Title: Isokinetic Exercise Combined With Blood Flow Restriction: High-Load Vs Low-Load Training : A Randomized Controlled Trial in Post-ACL Reconstruction Populations
Brief Title: Isokinetic Exercise Combined With Blood Flow Restriction: High-Load Vs Low-Load Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GulfMU
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: ACL Reconstruction; ACL Repair
Keywords: blood flow restriction training ACL; Blood flow restriction; ACL Rehab; ACLR; ACL Reconstruction; BFR therapy anterior cruciate ligament reconstruction; BFR therapy ACLR; BFR Therapy; low-load versus high-load BFR knee rehabilitation; isokinetic strength training after ACL surgery; physiotherapy rehabilitation protocol ACL isokinetic BFR; Knee physiotherapy; ACL; ACL Isokinetic; ACLٍ Isokinetic
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL Reconstruction Population (Active Comparator)
  Interventions: Other: High Load Isokinetic Training with Blood Flow Restriction; Other: Low Load Isokinetic Training with Blood Flow Restriction
- Healthy Population (Active Comparator)
  Interventions: Other: High Load Isokinetic Training with Blood Flow Restriction; Other: Low Load Isokinetic Training with Blood Flow Restriction

INTERVENTIONS:
Other: High Load Isokinetic Training with Blood Flow Restriction — High Load strength training that was administered through the use of an isokinetic device, and not conventional strength training equipment, combined with blood flow restriction.
  Other Names: High Load strength training; High Load Isokinetic training; Blood Flow Restriction; BFR
Other: Low Load Isokinetic Training with Blood Flow Restriction — Low Load strength training that was administered through the use of an isokinetic device, and not conventional strength training equipment, combined with blood flow restriction.
  Other Names: Low Load strength training; Low Load Isokinetic training; Blood Flow Restriction; BFR

SUMMARY:
The goal of this clinical trial is to see which type of strengthening exercise with a tight band (blood flow restriction) helps people recover better after ACL reconstruction. The study includes adults after ACL surgery who are doing physiotherapy to rebuild thigh muscle strength and knee function.

The main questions are:

* Does heavy strengthening with blood flow restriction improve thigh strength, knee function, and daily activities more than light strengthening with blood flow restriction after ACL surgery?
* Can light strengthening with blood flow restriction give similar benefits to heavy strengthening while putting less strain on the knee?

Researchers will compare a heavy-exercise program plus blood flow restriction to a light-exercise program plus blood flow restriction to see which gives better strength and functional improvements.

Participants will:

* Come for supervised physiotherapy sessions and do knee exercises on a machine, using either heavy or light loads while a cuff on the thigh gently squeezes to reduce blood flow.
* Have their leg strength, and knee questionnaires checked several times during the study.

DETAILED DESCRIPTION:
This clinical trial is testing two different ways of doing strength training with a tight leg cuff (blood flow restriction) during rehabilitation after ACL reconstruction. The aim is to find out which program helps people rebuild thigh muscle strength and knee function more effectively, while still keeping the knee joint safe after surgery.

Study purpose and questions After ACL reconstruction, many people lose muscle size and strength in the front of the thigh, which can slow down recovery and delay return to sport or full activity. Blood flow restriction training allows people to train with lighter weights but still gain strength and muscle, which may be useful when heavy loads are not yet safe.

The main questions are:

* Does a heavy-load isokinetic exercise program with blood flow restriction improve thigh strength, knee function, and patient-reported outcomes more than a low-load isokinetic program with blood flow restriction?
* Can low-load isokinetic exercise with blood flow restriction provide similar benefits in strength and function, while placing less stress on the healing knee joint? Who will take part The study will include adults who have had ACL reconstruction and are in the strengthening phase of their rehabilitation. Participants will typically be active people, cleared by their surgeon and physiotherapist to start moderate to high resistance training, with no serious heart, blood vessel, or bleeding problems that would make blood flow restriction unsafe.

What happens in the study Participants will be randomly assigned to one of two groups so that each person has an equal chance of being in either group.

* One group will do heavy-load isokinetic knee exercises with a blood flow restriction cuff on the thigh.
* The other group will do low-load isokinetic knee exercises with the same type of cuff and similar exercise schedule.

Both groups will:

* Attend supervised physiotherapy sessions several times per week for around 3-4 months.
* Perform knee extension and flexion exercises on an isokinetic machine, where the speed of movement is controlled and resistance adjusts through the range of motion.
* Wear a wide cuff around the upper thigh, which is inflated to a set pressure to partially reduce blood flow out of the leg during sets, then deflated during rest periods.

The physiotherapist will adjust the load (heavy or light), cuff pressure, and number of sets and repetitions according to a fixed protocol so that each participant trains safely and progressively over time.

Measurements and outcomes

Participants will be tested at the start of the study and at follow-up visits (for example, after several weeks and at the end of the program). The main outcome is peak quadriceps strength measured on an isokinetic dynamometer. Other outcomes may include:

* Rate of torque development (how quickly the muscle can produce force).
* Functional tests such as hop tests, walking or stair tests, and timed tasks.
* Patient questionnaires about knee symptoms, daily activities, sports function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

For ACLR group:

•Isolated unilateral ACL reconstruction 8-16 weeks post-surgery with medical clearance for moderate to high resistance training.

For control group(healthy population):

* Healthy adults with no musculoskeletal pathology.

Exclusion Criteria:

* History of cardiovascular or metabolic diseases
* Deep vein thrombosis
* Coagulopathy
* Hypertension
* Skin lesions or infections at the site of BFR cuff administration
* Neuromuscular disorders
* Non-clearance from the surgeon or physiotherapist or resistance training.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength | Outcome measures will be measured at baseline(week 0), mid-intervention(week 3) and post-intervention(week 6)
  Muscle strength will be measured using Biodex System 4 Pro for concentric quadriceps and hamstring strength at 60°/s and eccentric quadriceps at 60°/s.
  Recorded parameters: peak torque(Nm/kg), total work(J), and average power(W).
Muscle Girth | Outcome measures will be measured at baseline(week 0), mid-intervention(week 3) and post-intervention(week 6)
  Muscle girth will be measured by measuring the mid-thigh circumference using an inch tape at 15cm above the superior border of the patella. The mean of two readings will be recorded

SECONDARY OUTCOMES:
Pain Reduction | Outcome measures will be measured at baseline(week 0), mid-intervention(week 3) and post-intervention(week 6)
  Pain will be evaluated using the Numeric Pain Rating Scale(0-10). This refers to the pain the patient experiences in their operated knee and will observe how it changes with administration of the intervention(s).
  Scale: 0-10 Minimum value: 0 Maximum value: 10 Higher is worse(more pain). Lower is better(less pain)
Blood Flow | Outcome measures will be measured at baseline(week 0), mid-intervention(week 3) and post-intervention(week 6)
  The blood flow to the affected knee will be assessed by using infrared thermography(IRT) using standardized imaging protocols(room temperature 20-24°C, 40-60% humidity).
Tolerability and Perception of the Intervention(s) | Outcome measures will be measured at baseline(week 0), mid-intervention(week 3) and post-intervention(week 6)
  This will be recorded using a Likert-type questionnaire focusing on comfort, tightness, and willingness to repeat the intervention.
  Minimum value: 0 Maximum value: 10 Higher scores mean a better outcome. Lower scores mean a worse outcome.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reid D. Predicting maximal strength of quadriceps from submaximal performance in individuals with knee joint osteoarthritis. Arthritis Care & Research. 2011; doi:10.1002/ACR.20368
- [Background] de Deus Passos M, da Rocha AF. Evaluation of infrared thermography with a portable camera as a diagnostic tool for peripheral arterial disease of the lower limbs compared with color Doppler ultrasonography. Arch Med Sci Atheroscler Dis. 2022 Aug 8;7:e66-e72
- [Background] Côrte AC, Pedrinelli A, Marttos A, Souza IFG, Grava J, José Hernandez A. Infrared thermography study as a complementary method of screening and prevention of muscle injuries: pilot study. BMJ Open Sport & Exercise Medicine. 2019
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856
- [Background] Cvjetkovic DD, Bijeljac S, Palija S, Talic G, Radulovic TN, Kosanovic MG, Manojlovic S. Isokinetic Testing in Evaluation Rehabilitation Outcome After ACL Reconstruction. Med Arch. 2015 Feb;69(1):21-3. doi: 10.5455/medarh.2015.69.21-23
- [Background] Gopinatth V, Garcia JR, Reid IK, Knapik DM, Verma NN, Chahla J. Blood Flow Restriction Enhances Recovery After Anterior Cruciate Ligament Reconstruction: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Arthroscopy. 2025 Apr;41(4):1048-1060
- [Background] Lin Q, Zhang Y, Qin J, Wu F. Effects of Low-Load Blood Flow Restriction Training on Muscle Volume After Anterior Cruciate Ligament Reconstruction: A Systematic Review and Meta-analysis. Orthop J Sports Med. 2024 Dec 13;12(12):23259671241301731
- [Background] Koc B, Jansen E, de Jong O, et al. Qualitative Evaluation of Patient Experiences with Low-Load Blood Flow Restriction and Heavy-Load Resistance Training Post-ACL Reconstruction. IJSPT. 2025;20(10):1479-1488
- [Background] Koc BB, Truyens A, Heymans MJLF, Jansen EJP, Schotanus MGM. Effect of Low-Load Blood Flow Restriction Training After Anterior Cruciate Ligament Reconstruction: A Systematic Review. Int J Sports Phys Ther. 2022 Apr 1;17(3):334-346
- [Background] Moletta C, Kuenze CM, Morgan K, Coiner DR, Jacobson TA, Schmitz KH, Zajac NN, Boumerhi JS, Grindstaff TL. Hamstrings volumetric adaptations to a four-week Nordic hamstring exercise protocol in individuals with ACL reconstruction: a preliminary case series. Int J Sports Phys Ther. 2025 Sep 1;20(5):801-814
- [Background] Mengis N, Höher J, Ellermann A, Eberle C, Hartner C, Keller M, Rippke JN, Sprenger N, Stein T, Stoffels T, Egloff C, Niederer D. A Guideline for Validated Return-to-Sport Testing in Everyday Clinical Practice: A Focused Review on the Validity, Reliability, and Feasibility of Tests Estimating the Risk of Reinjury After ACL Reconstruction. Orthop J Sports Med. 2025 May 5;13(5):23259671251317208
- [Background] Hiemstra LA, Webber S, MacDonald PB, Kriellaars DJ. Contralateral limb strength deficits after anterior cruciate ligament reconstruction using a hamstring tendon graft. Clin Biomech (Bristol). 2007 Jun;22(5):543-50
- [Background] Kuenze C, Hart JM. Quadriceps strength thresholds and patient-reported function after anterior cruciate ligament reconstruction: a systematic review. J Sport Rehabil. 2023 Jun 1;32(5):458-468. doi: 10.1123/jsr.2022-0362
- [Background] Schwery NA, Kiely MT, Larson CM, Wulf CA, Heikes CS, Hess RW, Giveans MR, Solie BS, Doney CP. Quadriceps strength following anterior cruciate ligament reconstruction: normative values based on sex, graft type and meniscal status at 3, 6 & 9 months. Int J Sports Phys Ther. 2022 Apr 1;17(3):434-444
- [Background] Liao LR, Ng GYF, Jones AY, Lee LK, Leung HK, Ng SSM. Predicting maximal strength of quadriceps from submaximal performance in individuals with knee joint osteoarthritis. J Orthop Sports Phys Ther. 2015;45(5):408-414
- [Background] Nascimento DCN, Rolnick N, Sousa Neto IV, Severin R, Beal FLR. A useful blood flow restriction training risk stratification for exercise and rehabilitation. Front Physiol. 2022 Mar 11;13:808622
- [Background] Welsh JJ, Robinson DM, Dankel SJ. A systematic review examining blood flow restriction in combination with isokinetic resistance exercise. J Trainology. 2024;13(1):3-11
- [Background] Hughes L, Patterson SD, Haddad F, Rosenblatt B, Gissane C, McCarthy D, Clarke T, Ferris G, Dawes J, Paton B. Examination of the comfort and pain experienced with blood flow restriction training during post-surgery rehabilitation of anterior cruciate ligament reconstruction patients: A UK National Health Service trial. Phys Ther Sport. 2019 Sep;39:90-98
- [Background] Rolnick N, Kimbrell K, Cerqueira MS, Weatherford B, Brandner C. Perceived barriers to blood flow restriction training. Front Rehabil Sci. 2021 Jul 8;2:697082
- [Background] Farooq U, Cheema MY, Imran M, Gulzar M. Acute and chronic blood flow restriction resistance training: mechanisms and applications in sports. J Exerc Sci Fit. 2025;23(2):279-288
- [Background] Büyüklüoğlu G, Akinoğlu B, Günaydin H, Küçük İ, Örsçelik A, Kocahan T. Isokinetic exercise combined with blood flow restriction (BFR) may produce a greater change in the angle of peak torque. Med Sport. 2025;78(1):18-22
- [Background] Kubosch EJ, Izadi M, Wawrzyniak N, Hedtmann K, Pässler V, Rolvien T, von der Heide D, Lutter C, Fehér D, Engelhardt M. Blood flow restriction training for hamstring muscle strength after anterior cruciate ligament reconstruction: a randomized controlled trial. Knee. 2024 Aug;41:2444-2452
- [Background] Kwon S, Bae KC, Yon CJ, Kim DH. Current narrative review-application of blood flow restriction exercise in clinical knee problems. Medicina (Kaunas). 2025 Jul 30;61(8):1377
- [Background] Su C, Zhang Z, Liang B, Zhou S, Long X. Effects of blood flow restriction combined with high-load training on muscle strength and sports performance in athletes: a systematic review and meta-analysis. Front Physiol. 2025;16:1603568
- [Background] Piskin NE, Aktug ZB, Kara M, Yavuz G, Ozturk GT, Ibis S, Aka H. The effect of blood flow restriction training on isokinetic strength, muscle thickness and athletic performance. J Musculoskelet Neuronal Interact. 2025;25(2):208-218
- [Background] Chang H, Yan J, Lu G, Chen B, Zhang J. Muscle strength adaptation between high-load resistance training versus low-load blood flow restriction training with different cuff pressure characteristics: a systematic review and meta-analysis. Front Physiol. 2023 Aug 25;14:1244292
- [Background] Colombo V, Valenčič T, Steiner K, Škarabot J, Folland J, O'Sullivan O, Kluzek S. Comparison of blood flow restriction interventions to standard rehabilitation after an anterior cruciate ligament injury: a systematic review. Am J Sports Med. 2024 Apr 9;52(14):3641-3650